CLINICAL TRIAL: NCT03933410
Title: A Phase 2, Open-label Study to Evaluate the Efficacy and Safety of KB195 in Subjects With A Urea Cycle Disorder With Inadequate Control on Standard of Care
Brief Title: UNLOCKED: A Phase 2, Open-label Trial With KB195 in Subjects With a Urea Cycle Disorder
Acronym: UNLOCKED
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Kaleido Biosciences, Inc. closed the K020-218 trial due to business reasons, and not due to any safety concerns.
Sponsor: Kaleido Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K020-218
Record Dates: First submitted 2019-04-29; First posted 2019-05-01 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Urea Cycle Disorder
Keywords: Microbiome; Elevated Ammonia; Disorder of the Urea Cycle Metabolism; Urea Cycle Disorder; KB195; Kaleido; UNLOCKED; Ornithine Transcarbamylase Deficiency (OTC); Carbamoyl Phosphatase Synthetase 1 (CPS1); Argininosuccinic Acid Synthetase (ASS1); Argininosuccinic Acid Lyase (ASL); Arginase (ARG 1); N-acetyl Glutamate Synthetase (NAGS); Ornithine Translocase (ORNT1); Microbiome Metabolic Therapy (MMT); Glycan; Nitrogen Binding Therapy (NBT); Quality of Life; Oligosaccharide; Pediatric; Glutamine
MeSH Terms: conditions — Urea Cycle Disorders, Inborn; Ornithine Carbamoyltransferase Deficiency Disease

STUDY DESIGN:
Intervention Model Description: K020-218 is a single arm, open-label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- KB195 (Experimental): KB195 is a novel glycan
  Interventions: Drug: KB195

INTERVENTIONS:
Drug: KB195 — KB195 is a novel glycan

SUMMARY:
UNLOCKED: A Phase 2 Trial to Evaluate the Efficacy and Safety of KB195 in Subjects with a Urea Cycle Disorder with Inadequate Control on Standard of Care

DETAILED DESCRIPTION:
We expect the trial to enroll approximately 24 Urea Cycle Disorder (UCD) patients on standard of care with elevated ammonia levels. The planned treatment duration is eight weeks, with a primary endpoint of proportion of subjects who achieve a ≥15% reduction from baseline in fasting ammonia at the end of treatment. Patients will also be followed for safety and tolerability. This clinical trial is intended to allow us to evaluate efficacy of KB195 in reducing ammonia in UCD patients.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed informed consent and willing to comply with protocol-specified procedures.
* Has any confirmed UCD other than N-acetyl glutamatesynthase (NAGS) deficiency.
* Is male or female, 12 to 70 years of age (inclusive)
* If ≥ 18 years old, has a BMI ≥20.0 and < 40.0 kg/m2. If < 18 years old, has a BMI between 5th percentile and 95th percentile and weight greater than 5th percentile according to age, sex and regionally appropriate growth chart
* Has evidence of poorly controlled disease on the current standard of care (SOC)
* If NBT is part of SOC, is on a stable dose and regimen for at least 4 weeks before Screening and the dose is expected to remain stable during the study
* Is willing to maintain a stable diet throughout the course of study and is willing to continue usual exercise routine.
* If taking probiotics or prebiotics, is on a stable dose regimen for at least 4 weeks before Screening and the dose and regimen are expected to remain stable during the study
* Has a negative urine screen for drugs of abuse at Screening
* If male or female of child bearing potential, agree with use effective method of contraception for the duration of the study and 90 days after last dose of study product

Key Exclusion Criteria:

* Is at a high risk for metabolic decomposition.
* Has had a substantive change in diet or any other aspect of UCD management within 4 weeks before the Screening Visit
* Has used a systemic anti-infective within 4 weeks before the Screening Visit, or use is anticipated during the study
* Has been diagnosed with Citrullinemia Type II
* Is receiving any systemically administered immunosuppressant medication on a chronic basis
* Has changed the use of or dose of any drug or other compound to modulate GI motility within 4 weeks before the Screening Visit, or the use or dose is expected change during the course of the study
* Has a history of or active GI or liver disease
* Has a prior solid organ transplantation including liver transplantation, or is anticipated to receive a liver transplant during study participation
* Has used an investigational drug, product, or device within 30 days before the Screening Visit
* Has a contraindication, sensitivity, or known allergy to the study drug
* Is considered, in the opinion of the PI, to likely be a poor attendee or unlikely for any reason to be able to comply with the study drug procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who achieve a ≥15% reduction from baseline in fasting plasma ammonia at the end of treatment. | Day -1 to Day 55

SECONDARY OUTCOMES:
Proportion of subjects normalizing their fasting plasma ammonia concentrations from above the upper limit of normal at baseline to below the upper limit of normal at the end of treatment. | Day -1 to Day 55
Number of subjects experiencing adverse events (AEs) | Day -28 to Day 84
Number of subjects experiencing severe adverse events (SAEs) | Day -28 to Day 84
Change from baseline to end of treatment in Gastrointestinal Tolerability Questionnaire (GITQ) scores | Day -28 to Day 84
  Evaluate the effect of KB195 on self-report questionnaires including the Gastrointestinal Tolerability Questionnaire, an assessment of the frequency and severity of GI symptoms, e.g., gas, abdominal pain, calculated on a scale from 0 (None/Not applicable) to a maximum score of 60 (Severe/Much more than usual) for all questions
Change from baseline to end of treatment in Bristol Stool Scale (BSS) scoring. | Day -28 to Day 84
  Evaluate the effect of KB195 on self-report questionnaires including the Bristol Stool Scale, an assessment of stool consistency on a scale from 1 (separate hard lumps, like nuts, hard to pass) through 7 (watery, no solid pieces, entirely liquid)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Wingertzahn, PhD, Study Director — Kaleido Biosciences
Locations (19):
- United States (6):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of South Florida/ USF HEALTH, Tampa, Florida
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai-Clinical Research Unit, New York, New York
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
- Zentrum für Kinder- und Jugendmedizin Angelika-Lautenschläger-Klinik, Heidelberg, Germany
- Spain (4):
  - Hospital de Cruces, Barakaldo
  - Hosptial Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Virgen del Rocio, Seville
- Switzerland (2):
  - Inselpital, Universitaetsklinik fur Kinderheikunde, Bern
  - Inselpital, Universitätsklinik für Kinderheilkunde, Bern
- Department of Child Health and Diseases, Department of Nutrition and Metabolism Istanbul University, Istanbul, Turkey (Türkiye)
- United Kingdom (3):
  - Salford Royal Hospital, Salford, Greater Manchester
  - National Hospital for Neurology and Neurosurgery, London
  - Salford Royal NHS Foundation Trust, Salford